THE AFFECT OF AN ANTI-EMBOLISM STOCKING PROTOCOL ON THE DEVELOPMENT OF EARLY VENOUS THROMBOEMBOLIA IN PATIENTS WITH KNEE ARTROPLASTY

SHORT TITLE: THE AFFECT OF AN AES PROTOCOL

Specialist Nurse Ismail Furkan BAŞIBÜYÜK<sup>1</sup>

<sup>1</sup>Cukurova University Balcalı Hospital A Block 6<sup>th</sup> Floor Orthopedics and Traumatology Clinic Sarıcam/ADANA TURKEY, Tel: 0531-959-95-43, Email: <u>ifurkan01@gmail.com</u>, ORCID No: 0000-0003-3480-769X

Assoc. Prof. Dr. Sevilay ERDEN<sup>2</sup> [Corresponding Author]

<sup>2</sup>Cukurova University Faculty of Health Sciences Department of Surgery Sarıcam/ADANA TURKEY, Tel: 0539-323-18-72, Email: <a href="mailto:sevilaygil@gmail.com">sevilaygil@gmail.com</a>, ORCID No: 0000-0002-6519-864X

**Acknowledgments:** We would like to thank the patients who contributed to the literature by agreeing to participate in the study, as well as all of the orthopedics clinic team members who helped with the study's implementation.

**Conflict if interest statement:** The authors declared no potential conflicts of interest with respect to the research, authorship, and/or publication of this article.

**Funding:** This study was supported by University Scientific Research Projects Coordination Unit under the project number "TYL-2019-12245".

## **Authorship Criteria**

Idea generation: IBF, SE

Literature review: IBF

Study design: IBF,SE

Data collection: IBF

Statistics//analysis: IBF,SE

Interpretation of the results: IBF,SE

Writing of the article: IBF,SE